CLINICAL TRIAL: NCT04262921
Title: Clinical Characterisation Protocol for Severe Emerging Infections
Brief Title: French COVID Cohort
Acronym: FrenchCOVID
Status: Active, not recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-05; 2020-A00256-33 (Registry Identifier: RCB ID)
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Coronavirus Infections
Keywords: Coronavirus; 2019-nCoV; COVID-19; SARS-CoV-2; Cohort
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool /rectal swab, respiratory samples (nose and throat swab, endotracheal aspirate, nasopharyngeal aspirate), samples from infected sites/sores, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious disease is the single biggest cause of death worldwide. New infectious agents, such as the SARS, MERS and other novel coronavirus, novel influenza viruses, viruses causing viral haemorrhagic fever (e.g. Ebola), and viruses that affect the central nervous system (CNS) such as TBEV & Nipah require investigation to understand pathogen biology and pathogenesis in the host. Even for known infections, resistance to antimicrobial therapies is widespread, and treatments to control potentially deleterious host responses are lacking.

In order to develop a mechanistic understanding of disease processes, such that risk factors for severe illness can be identified and treatments can be developed, it is necessary to understand pathogen characteristics associated with virulence, the replication dynamics and in-host evolution of the pathogen, the dynamics of the host response, the pharmacology of antimicrobial or host-directed therapies, the transmission dynamics, and factors underlying individual susceptibility.

The work proposed here may require sampling that will not immediately benefit the participants. It may also require analysis of the host genome, which may reveal other information about disease susceptibility or other aspects of health status.

ELIGIBILITY:
Inclusion Criteria:

- Any patient admitted to a health care facility, with an infection confirmed by SARS-CoV-2 (virologically confirmed diagnosis by PCR).

Non inclusion criteria:

* Subject deprived of freedom, subject under a legal protective measure
* Refusal by participant, parent or appropriate representative.

Exclusion Criteria:

- Confirmed diagnosis of another pathogen than SARS-CoV-2 and no indication or likelihood of co-infection with SARS-CoV-2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enrol eligible patients (children and adults) with confirmed infection with SARS-CoV-2. Recruitment of patients with Day 1 (enrolment) data is the priority.
  The patient's follow-up will be done strictly within the management adapted to his infection. No visits will be made specifically for research purposes. The organisation of convalescence visits is left to the discretion of each centre according to its post-hospitalisation patient follow-up procedures.
  Additional biological samples will be collected when samples are taken in the context of care in order to meet the research objectives, with the exception of certain blood samples for pharmacokinetic analyses.
Sampling Method: Probability Sample
Enrollment: 4415 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Clinical features | 18 months
  Describe the clinical features of the illness or syndrome (cardio-respiratory signs or symptoms, and laboratory results) and complications, and determinants of severity.
  Assessment daily for 15 days, then weekly until max 100 days, then 3 and 6 months.
Response to treatment | 18 months
  Describe the response to treatments (including supportive care and novel therapeutics) by clinical, biological, radiological and virological assessments.
  Assessment daily for 15 days, then weekly until max 100 days, then 3 and 6 months.
Pathogen replication, excretion and evolution, within the host | 18 months
  high-throughput sequencing of pathogen genomes obtained from respiratory tract, blood, urine, stool, CSF and other samples.
  Assessment on Day 1, Day 2, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 15 then weekly until max 100 days, then 3 and 6 months.
Immune host responses to infection and therapy | 18 months
  Characterise the innate and acquired immune responses, circulating levels of immune signalling molecules and gene expression profiling in peripheral blood.
  Assessment on Day 1, Day 2, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 15 then weekly until max 100 days, then 3 and 6 months.
Host genetic variants | Day 1
  Identify host genetic variants associated with disease progression or severity

CONTACTS AND LOCATIONS:
Overall Officials: Jade GHOSN, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (98):
- France (98):
  - CHG Agen, Agen
  - Centre Hospitalier Du Pays D'aix, Aix-en-Provence
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Annecy Genevois, Annecy
  - Hopital privé d'Antony, Antony
  - Hôpital de Mercy. CHR METZ-THIONVILLE, Ars-Laquenexy
  - Centre Hospitalier Henri Duffaut, Avignon
  - Chu Jean Minjoz, Besançon
  - Centre hospitalier de Béziers, Béziers
  - Hôpital Avicenne AP-HP, Bobigny
  - CHU Pellegrin, Bordeaux
  - CHU Ambroise Paré, Boulogne-Billancourt
  - Ch Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Chru Hopital Cavale Blanche, Brest
  - CHU Brest, Brest
  - Hospices civils de Lyon, Bron
  - CH Cahors, Cahors
  - Centre Hospitalier J.E Techer, Calais
  - Centre Hospitalier Andrée Rosemon, Cayenne
  - Chms Chambery Nh, Chambéry
  - Centre Hospitalier De Cholet, Cholet
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH Colmar - Hopital Pasteur, Colmar
  - Hôpital Louis Mourier, Colombes
  - Centre hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Dax, Dax
  - CHU Dijon Bourgogne, Dijon
  - CH Annecy Genevois, Épagny
  - CHU de Martinique, Fort de France
  - Hopital Raymond Poincare, Garches
  - CHU Grenoble, Grenoble
  - Grand Hopital de l'Est Francilien site Marne-la-Vallée, Jossigny
  - Chd Les Oudairies, La Roche-sur-Yon
  - Hôpital Universitaire Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier Universitaire de Lille, Lille
  - CHRU Lille, Hôpital Salengro, Lille
  - CHU de Lille, Lille
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Louis Raffalli, Manosque
  - Assistance publique hopitaux de Marseille, hopital Nord, Marseille
  - Hopital Européen, Marseille
  - Hôpital Conception, Marseille
  - Groupe Hospitalier Sud Ile De France, Melun
  - CH de Mont Marsan, Mont-de-Marsan
  - Groupe hospitalier du Havre, Montivilliers
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hopital Américain de Paris, Neuilly-sur-Seine
  - CHU de Nice, Nice
  - CHU Caremeau, Nîmes
  - APHP Bichat, Paris
  - APHP Tenon, Paris
  - CH Lariboisière, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hopital Cochin-CIC1417, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - La pitié salpetrière, Paris
  - Centre Hospitalier de Pau, Pau
  - CH de Perpignan, Perpignan
  - Centre Hospitalier de Périgueux, Périgueux
  - Hopital Lyon Sud-HCL, Pierre-Bénite
  - CHU de Pointe à Pitre, Pointe à Pitre
  - CHU de Poitiers, Poitiers
  - Ch Cornouaille, Quimper
  - Chu Reims, Reims
  - CHU Rennes Hopital Sud, Rennes
  - Hôpital Pontchaillou, Rennes
  - CHU Charles Nicole, Rouen
  - CHU Rouen Normandie, Rouen
  - CHU Réunion-Felix Guyon, Saint-Denis
  - CHU de Saint-Etienne, Saint-Etienne
  - Hopital d'instruction des armées Begin 69, Saint-Mandé
  - Centre hospitalier Louis Constant Fleming, Saint-Martin
  - Groupe Hospitalier Sud Réunion, Saint-Pierre
  - CH de Saintonge, Saintes
  - Centre Hospitalier de Soissons, Soissons
  - N.H.C. - Nouvel Hopital Civil, Strasbourg
  - Hopital Foch, Suresnes
  - CHR Metz-Thionville -Hopital Bel Air, Thionville
  - Hopitaux du Leman, Thonon-les-Bains
  - Centre Hospitalier Universitaire de Rangueil, Toulouse
  - CHU de Toulouse, Toulouse
  - CHU Toulouse IUCT Institut Universitaire de Cancer de Toulouse, Toulouse
  - CHU Toulouse Larrey, Toulouse
  - Hôpital Gustave Dron, Tourcoing
  - Centre Hospitalier Régional Universitaire de Tours, Tours
  - CHRU de Tours, Tours
  - CHU Nancy, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reyes LF, Garcia-Gallo E, Murthy S, Fuentes YV, Serrano CC, Ibanez-Prada ED, Lee J, Rojek A, Citarella BW, Goncalves BP, Dunning J, Ratsep I, Vinan-Garces AE, Kartsonaki C, Rello J, Martin-Loeches I, Shankar-Hari M, Olliaro PL, Merson L; ISARIC Characterisation Group. Major adverse cardiovascular events (MACE) in patients with severe COVID-19 registered in the ISARIC WHO clinical characterization protocol: A prospective, multinational, observational study. J Crit Care. 2023 Oct;77:154318. doi: 10.1016/j.jcrc.2023.154318. Epub 2023 May 9. PMID 37167775
- [Derived] Matuozzo D, Talouarn E, Marchal A, Zhang P, Manry J, Seeleuthner Y, Zhang Y, Bolze A, Chaldebas M, Milisavljevic B, Gervais A, Bastard P, Asano T, Bizien L, Barzaghi F, Abolhassani H, Abou Tayoun A, Aiuti A, Alavi Darazam I, Allende LM, Alonso-Arias R, Arias AA, Aytekin G, Bergman P, Bondesan S, Bryceson YT, Bustos IG, Cabrera-Marante O, Carcel S, Carrera P, Casari G, Chaibi K, Colobran R, Condino-Neto A, Covill LE, Delmonte OM, El Zein L, Flores C, Gregersen PK, Gut M, Haerynck F, Halwani R, Hancerli S, Hammarstrom L, Hatipoglu N, Karbuz A, Keles S, Kyheng C, Leon-Lopez R, Franco JL, Mansouri D, Martinez-Picado J, Metin Akcan O, Migeotte I, Morange PE, Morelle G, Martin-Nalda A, Novelli G, Novelli A, Ozcelik T, Palabiyik F, Pan-Hammarstrom Q, de Diego RP, Planas-Serra L, Pleguezuelo DE, Prando C, Pujol A, Reyes LF, Riviere JG, Rodriguez-Gallego C, Rojas J, Rovere-Querini P, Schluter A, Shahrooei M, Sobh A, Soler-Palacin P, Tandjaoui-Lambiotte Y, Tipu I, Tresoldi C, Troya J, van de Beek D, Zatz M, Zawadzki P, Al-Muhsen SZ, Alosaimi MF, Alsohime FM, Baris-Feldman H, Butte MJ, Constantinescu SN, Cooper MA, Dalgard CL, Fellay J, Heath JR, Lau YL, Lifton RP, Maniatis T, Mogensen TH, von Bernuth H, Lermine A, Vidaud M, Boland A, Deleuze JF, Nussbaum R, Kahn-Kirby A, Mentre F, Tubiana S, Gorochov G, Tubach F, Hausfater P; COVID Human Genetic Effort; COVIDeF Study Group; French COVID Cohort Study Group; CoV-Contact Cohort; COVID-STORM Clinicians; COVID Clinicians; Orchestra Working Group; Amsterdam UMC Covid-19 Biobank; NIAID-USUHS COVID Study Group; Meyts I, Zhang SY, Puel A, Notarangelo LD, Boisson-Dupuis S, Su HC, Boisson B, Jouanguy E, Casanova JL, Zhang Q, Abel L, Cobat A. Rare predicted loss-of-function variants of type I IFN immunity genes are associated with life-threatening COVID-19. Genome Med. 2023 Apr 5;15(1):22. doi: 10.1186/s13073-023-01173-8. PMID 37020259
- [Derived] Hocini H, Wiedemann A, Blengio F, Lefebvre C, Cervantes-Gonzalez M, Foucat E, Tisserand P, Surenaud M, Coleon S, Prague M, Guillaumat L, Krief C, Fenwick C, Laouenan C, Bouadma L, Ghosn J, Pantaleo G, Thiebaut R; French COVID cohort study group; Levy Y. Neutrophil Activation and Immune Thrombosis Profiles Persist in Convalescent COVID-19. J Clin Immunol. 2023 Jul;43(5):882-893. doi: 10.1007/s10875-023-01459-x. Epub 2023 Mar 21. PMID 36943669
- [Derived] Legrand M, Fong N, Laouenan C, Ghosn J, Thill B, Faure K, Garot D, Goujard C, Curlier E, Resche-Rigon M, Rossignol P, Pirracchio R. Risk factors of long term symptoms and outcomes among patients discharged after covid-19: prospective, multicentre observational study. BMJ Med. 2022 Jun 17;1(1):e000093. doi: 10.1136/bmjmed-2021-000093. eCollection 2022. PMID 36936553
- [Derived] Baruch J, Rojek A, Kartsonaki C, Vijayaraghavan BKT, Goncalves BP, Pritchard MG, Merson L, Dunning J, Hall M, Sigfrid L, Citarella BW, Murthy S, Yeabah TO, Olliaro P; ISARIC Clinical Characterisation Group. Symptom-based case definitions for COVID-19: Time and geographical variations for detection at hospital admission among 260,000 patients. Influenza Other Respir Viruses. 2022 Nov;16(6):1040-1050. doi: 10.1111/irv.13039. Epub 2022 Sep 5. PMID 36825252
- [Derived] Marwali EM, Kekalih A, Yuliarto S, Wati DK, Rayhan M, Valerie IC, Cho HJ, Jassat W, Blumberg L, Masha M, Semple C, Swann OV, Kohns Vasconcelos M, Popielska J, Murthy S, Fowler RA, Guerguerian AM, Streinu-Cercel A, Pathmanathan MD, Rojek A, Kartsonaki C, Goncalves BP, Citarella BW, Merson L, Olliaro PL, Dalton HJ; International Severe Acute Respiratory and emerging Infection Consortium (ISARIC) Clinical Characterization Group Investigators. Paediatric COVID-19 mortality: a database analysis of the impact of health resource disparity. BMJ Paediatr Open. 2022 Oct;6(1):e001657. doi: 10.1136/bmjpo-2022-001657. PMID 36645791
- [Derived] Garcia L, Woudenberg T, Rosado J, Dyer AH, Donnadieu F, Planas D, Bruel T, Schwartz O, Prazuck T, Velay A, Fafi-Kremer S, Batten I, Reddy C, Connolly E, McElheron M, Kennelly SP, Bourke NM, White MT, Pelleau S. Kinetics of the SARS-CoV-2 Antibody Avidity Response Following Infection and Vaccination. Viruses. 2022 Jul 8;14(7):1491. doi: 10.3390/v14071491. PMID 35891471
- [Derived] Gault N, Esposito-Farese M, Revest M, Inamo J, Cabie A, Polard E, Hulot JS, Ghosn J, Chirouze C, Deconinck L, Diehl JL, Poissy J, Epaulard O, Lefevre B, Piroth L, De Montmollin E, Oziol E, Etienne M, Laouenan C, Rossignol P, Costagliola D, Vidal-Petiot E; French-Covid cohort investigators, study group. Chronic use of renin-angiotensin-aldosterone system blockers and mortality in COVID-19: A multicenter prospective cohort and literature review. Fundam Clin Pharmacol. 2021 Dec;35(6):1141-1158. doi: 10.1111/fcp.12683. Epub 2021 May 16. PMID 33876439
- [Derived] Buetti N, Wicky PH, Le Hingrat Q, Ruckly S, Mazzuchelli T, Loiodice A, Trimboli P, Forni Ogna V, de Montmollin E, Bernasconi E, Visseaux B, Timsit JF. SARS-CoV-2 detection in the lower respiratory tract of invasively ventilated ARDS patients. Crit Care. 2020 Oct 16;24(1):610. doi: 10.1186/s13054-020-03323-5. PMID 33066801
- [Derived] Bouadma L, Wiedemann A, Patrier J, Surenaud M, Wicky PH, Foucat E, Diehl JL, Hejblum BP, Sinnah F, de Montmollin E, Lacabaratz C, Thiebaut R, Timsit JF, Levy Y. Immune Alterations in a Patient with SARS-CoV-2-Related Acute Respiratory Distress Syndrome. J Clin Immunol. 2020 Nov;40(8):1082-1092. doi: 10.1007/s10875-020-00839-x. Epub 2020 Aug 22. PMID 32829467